CLINICAL TRIAL: NCT01148537
Title: A Randomized, Double-blind, Placebo- & Positive-Controlled, Parallel Group, Dose Escalating Study to Evaluate the Effect of Buprenorphine Delivered by Buprenorphine Transdermal System at 10- and 40-mg Dose Levels on QT Intervals in Healthy Adult Volunteers
Brief Title: The Effect of Buprenorphine Delivered by Buprenorphine Transdermal System (BTDS) on QT Intervals in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUP1011
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Results first posted 2010-09-28 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy subjects; Opioid; Transdermal
MeSH Terms: interventions — Buprenorphine; Moxifloxacin; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- BTDS (Experimental): Buprenorphine transdermal patches 5, 10, 20, and 2 * 20 mcg/h.
  Interventions: Drug: Buprenorphine transdermal patch
- Placebo TDS (Placebo Comparator): Matching placebo transdermal patches 5, 10, 20 and 2 * 20.
  Interventions: Drug: Matching placebo transdermal patch
- Moxifloxacin (Active Comparator): Moxifloxacin hydrochloride 400 mg tablets
  Interventions: Drug: Avelox (moxifloxacin hydrochloride) tablet

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 5, 10, 20, and 2 * 20 mcg/h.
  Other Names: Butrans™
  Arms: BTDS
Drug: Matching placebo transdermal patch — Placebo transdermal patch to match BTDS 5, 10, 20, and 2 * 20.
  Arms: Placebo TDS
Drug: Avelox (moxifloxacin hydrochloride) tablet — Moxifloxacin 400 mg tablet; 1 tablet taken orally on days 6 and 13
  Other Names: Avelox
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to examine the effect of buprenorphine on QT interval corrected for heart rate (QTc) in healthy subjects.

DETAILED DESCRIPTION:
Drugs in this opioid class have been associated with prolonging QT interval/QT interval corrected for heart rate (QTc).

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 55 years of age, inclusive.
* Body weight ranging from 50 to 100 kilograms (kg) and a body mass index (BMI) ≤ 30 kg/m2.
* Healthy as determined by unremarkable medical history, physical examination, vital signs, laboratory evaluations, electrocardiogram (ECG), and a 24-hour screening ECG telemetry.
* Willing to refrain from strenuous exercise or contact sports during the study.
* Female subjects must be surgically sterile or at least 2 years postmenopausal, or using an effective contraceptive method (intrauterine device, hormonal contraceptive, or double-barrier method).

Exclusion Criteria:

* Any clinically significant illness during the 30 days prior to randomization.
* Any history of allergy to buprenorphine, any excipient of BTDS, opioids, psychotropic or hypnotic drugs, and/or moxifloxacin or any member of the quinolone class of drugs.
* A clinically significant history of allergic reaction to wound dressings or bandages.
* Any medical or surgical conditions which might interfere with drug absorption (transdermal or gastrointestinal), distribution, metabolism, or excretion.
* Abnormalities on physical examination, vital signs, ECG, or clinical laboratory values, unless those abnormalities are judged to be clinically insignificant by the Investigator.
* Any cardiovascular disorders, including hypertension.
* Oxygen saturation (SpO2) ≤ 94% as measured by pulse oximetry.
* Any personal or family history of prolonged QT interval or disorders of cardiac rhythm.
* Abnormal cardiac condition denoted by any of the following:
* QT interval ≥ 450 milliseconds (msec).
* PR interval > 240 msec or ≤ 110 msec.
* Evidence of second- or third-degree atrioventricular (AV) block.
* Pathological Q-waves (defined as Q-wave > 40 msec or depth > 0.5 mV).
* Evidence of ventricular preexcitation, complete left bundle branch block, right bundle branch block (RBBB), or incomplete RBBB.
* A resting heart rate outside the range of 50 to 85 beats per minute (bpm).

Other protocol-specific exclusion/inclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2004-07; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP, Clinics, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 02-Jul-2004 (first patient first visit) to 16-Dec-2004 (last patient last visit) at 1 site in the US (Austin, TX.)
Pre-assignment Details: During the initial screening visit, subjects were assessed for study eligibility through medical history, physical examination, vital signs, oxygen saturation, conventional 12-lead ECG, and laboratory tests. The investigator at the site examined the ECG telemetry to determine the subjects' eligibility.
Groups:
- BTDS: Buprenorphine transdermal patches 5, 10, 20, and 2 * 20 mcg/h. Randomization was from predose on day 1 to predose on day 14. There were 3 treatment groups: BTDS, placebo, and moxifloxacin as the positive control. The treatment groups between placebo and BTDS were double-blinded. Moxifloxacin treatment was open label to subjects, to the investigator, and the staff at the study site.
  BTDS or placebo TDS was applied on day 1 for 3 days (BTDS 5), on day 4 for 3 days (BTDS 10), on day 7 for 3 days (BTDS 20), and on day 10 for 4 days (2 * BTDS 20). On day 6 and day 13, subjects in the positive control group received one 400 mg tablet of moxifloxacin.
- Placebo: Matching placebo transdermal patches.
- Moxifloxacin: Positive control: One 400 mg moxifloxacin tablet (Avelox®) by mouth on days 6 and 13
Period: Overall Study
Arm/Group | BTDS | Placebo | Moxifloxacin
Started | 44 | 44 | 44
Completed | 41 | 44 | 41
Not Completed | 3 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Adverse Event | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BTDS | Placebo | Moxifloxacin | Total
Number analyzed (Participants) | 44 | 44 | 44 | 132
Age Continuous [Mean (Standard Deviation); unit: years] | 30.8 (9.46) | 34.1 (10.7) | 28.8 (9.69) | 31.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 23 | 68
  Male | 22 | 21 | 21 | 64

OUTCOME MEASURES:

1. Primary Outcome: The Comparison of BTDS to Placebo Transdermal System (TDS): the Average Difference From Baseline Using QT Corrected From Within-subject Data (QTci) on Day 13
Description: Observed time from start of the QRS complex to end of the T wave (QT), and the time between the 2 R waves (RR) data for each of 4 electrocardiographs (ECGs) over an approximate 10-minute interval at each nominal time point. The average QT and QTc data over the 2 pretreatment days were used as the baseline.
  Observed time from start of the QRS complex to end of the T wave (QT); interval corrected for heart rate (QTc) msec; interval corrected from within-subject data (QTci) msec.
Time Frame: Baseline to Day 13
Population: The full analysis population for ECGs (N = 131) was defined as all subjects who received at least 1 dose of study drug and had at least 1 postdose digital QT/QTc evaluation.
  For the comparison of BTDS to placebo (N = 88), the subjects randomized to moxifloxacin were excluded.
Measure: Least Squares Mean (Standard Deviation); unit: QTci (msec)
Arm/Group | BTDS | Placebo
Number analyzed (Participants) | 44 | 44
QTci (msec) | 4.20 (7.44) | -1.71 (6.92)
Statistical Analysis 1: Comparison: BTDS vs Placebo; Test type: Superiority or Other; p < .001, ANCOVA; ANCOVA model with baseline QTci as a covariate and with sex and treatment as effects in the model; Mean Difference (Final Values) = 5.91, 90% CI 2-sided [3.4 to 8.4]

2. Secondary Outcome: The Average Differences Between BTDS vs Placebo From Baseline by Interval Corrected From Within-subject Data (QTci) on Day 6
Description: QT and RR data were determined for each of 4 ECGs over an approximate 10-minute interval at each nominal time point. The average QT and QTc data from the replicate ECGs at each nominal time point were calculated. The average QT and QTc data over the 2 pretreatment days were used as the baseline QT and QTc values.
  Observed time from start of the QRS complex to end of the T wave (QT); interval corrected for heart rate (QTc) msec; interval corrected from within-subject data (QTci) msec.
Time Frame: Baseline to Day 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: QTci (msec)
Arm/Group | BTDS | Placebo
Number analyzed (Participants) | 44 | 44
QTci (msec) | -1.06 (6.17) | -1.46 (6.69)
Statistical Analysis 1: Comparison: BTDS vs Placebo; Test type: Superiority or Other; p = .770, ANCOVA; Mean Difference (Final Values) = 0.39, 90% CI 2-sided [-1.8 to 2.6] — For the comparison of BTDS to placebo, the subjects randomized to moxifloxacin were excluded

3. Primary Outcome: The Comparison of Moxifloxacin to Placebo Transdermal System (TDS): the Average Difference From Baseline Using QT Interval Corrected From Within-subject Data (QTci) on Day 13
Description: Observed time from start of the QRS complex to end of the T wave (QT), and the time between the 2 R waves (RR) data for each of 4 electrocardiographs (ECGs) over an approximate 10-minute interval at each nominal time point. The average QT and QTc data over the 2 pretreatment days were used as the baseline QT and QTc values.
  Observed time from start of the QRS complex to end of the T wave (QT); interval corrected for heart rate (QTc) msec; interval corrected from within-subject data (QTci) msec.
Time Frame: Baseline to Day 13
Population: The full analysis population for ECGs (N = 131) was defined as all subjects who received at least 1 dose of study drug and had at least 1 postdose digital QT/QTc evaluation.
  For the comparison of moxifloxacin to placebo (N=88), the subjects randomized to BTDS were excluded.
Measure: Least Squares Mean (Standard Deviation); unit: QTci (msec)
Groups:
- Moxifloxacin: Positive Control: One 400 mg moxifloxacin tablet by mouth on days 6 and 13.
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 44 | 44
QTci (msec) | 4.17 (7.22) | -1.69 (6.92)
Statistical Analysis 1: Comparison: Moxifloxacin vs Placebo; Day 13 analysis; Test type: Superiority or Other; p < .001, ANCOVA; ANCOVA model with baseline QTci as a covariate and with sex and treatment as effects in the model; Mean Difference (Final Values) = 5.86, 90% CI 2-sided [3.3 to 8.4]

4. Secondary Outcome: The Average Differences Between Moxifloxacin vs Placebo From Baseline by Interval Corrected From Within-subject Data (QTci) on Day 6
Description: as for outcome 2
Time Frame: Baseline to Day 6
Population: The full analysis population for ECGs (N = 131) was defined as all subjects who received at least 1 dose of study drug and had at least 1 postdose digital QT/QTc evaluation
  For the comparison of moxifloxacin to placebo (N = 88), the subjects randomized to BTDS were excluded.
Measure: Least Squares Mean (Standard Deviation); unit: QTci (msec)
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 44 | 44
QTci (msec) | 6.26 (6.11) | -1.38 (6.69)
Statistical Analysis 1: Comparison: Moxifloxacin vs Placebo; Test type: Superiority or Other; p < .001, ANCOVA; ANCOVA model with average baseline as a covariate, and with gender and treatment as main effects; Mean Difference (Final Values) = 7.64, 90% CI 2-sided [5.4 to 9.9]

5. Secondary Outcome: The Average Differences From Baseline Between BTDS and Placebo by Bazett Corrected QT Interval (QTcB) on Day 6 and Day 13
Description: QT and RR data were determined for each of 4 ECGs over an approximate 10-minute interval at each nominal time point. The average QT and QTc (QT interval corrected for heart rate) data from the replicate ECGs at each nominal time point were calculated. The average QT and QTc data over the 2 pretreatment days were used as the baseline QT and QTc values.
  Observed time from start of the QRS complex to end of the T wave (QT); interval corrected for heart rate (QTc) msec; interval corrected by Bazett's method (QTcB) msec.
Time Frame: Baseline to Day 6 and Day 13
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: QTcB (msec)
Arm/Group | BTDS | Placebo
Number analyzed (Participants) | 44 | 44
QTcB (msec)
  QTcB Day 6 | -0.37 (7.18) | -0.24 (8.15)
  QTcB Day 13 | 6.31 (8.73) | -0.86 (8.49)
Statistical Analysis 1: Comparison: BTDS vs Placebo; Day 6 analysis; Test type: Superiority or Other; p = .936, ANCOVA; Mean Difference (Final Values) = -0.13, 90% CI 2-sided [-2.9 to 2.6]
Statistical Analysis 2: Comparison: BTDS vs Placebo; Day 13 analysis; Test type: Superiority or Other; p < .001, ANCOVA; Mean Difference (Final Values) = 7.16, 90% CI 2-sided [4.2 to 10.1]

6. Secondary Outcome: The Average Differences From Baseline Between Moxifloxacin and Placebo of Bazett Corrected QT Interval (QTcB) on Day 6 and Day 13
Description: QT and RR data were determined for each of 4 ECGs over an approximate 10-minute interval at each nominal time point. The average QT and QTc data from the replicate ECGs at each nominal time point were calculated. The average QT and QTc data over the 2 pretreatment days were used as the baseline QT and QTc values.
  Observed time from start of the QRS complex to end of the T wave (QT); interval corrected for heart rate (QTc) msec; interval corrected by Bazett's method (QTcB) msec.
Time Frame: Baseline to Day 6 and Day 13
Population: as for outcome 3
Measure: Least Squares Mean (Standard Deviation); unit: QTcB (msec)
Groups:
- Mofloxacin: Positive Control: One 400 mg moxifloxacin tablet by mouth on days 6 and 13.
Arm/Group | Mofloxacin | Placebo
Number analyzed (Participants) | 44 | 44
QTcB (msec)
  QTcB Day 6 | 8.13 (6.92) | -0.09 (8.15)
  QTcB Day 13 | 6.55 (8.59) | -0.84 (8.49)
Statistical Analysis 1: Comparison: Mofloxacin vs Placebo; Day 6 analysis; Test type: Superiority or Other; p < .001, ANCOVA; Mean Difference (Final Values) = 8.23, 90% CI 2-sided [5.5 to 10.9]
Statistical Analysis 2: Comparison: Mofloxacin vs Placebo; Day 13 analysis; Test type: Superiority or Other; p < .001, ANCOVA; Mean Difference (Final Values) = 7.40, 90% CI 2-sided [4.3 to 10.5]

7. Secondary Outcome: The Average Differences From Baseline Between BTDS and Placebo by Fridericia's Corrected Interval (QTcF) on Day 6 and Day 13
Description: QT and RR data were determined for each of 4 ECGs over an approximate 10-minute interval at each nominal time point. The average QT and QTc (interval corrected for heart rate) data from the replicate ECGs at each nominal time point were calculated. The average QT and QTc data over the 2 pretreatment days were used as the baseline QT and QTc values.
  Observed time from start of the QRS complex to end of the T wave (QT); interval corrected for heart rate (QTc) msec; interval corrected by Fridericia's method (QTcF) msec.
Time Frame: Baseline to Day 6 and Day 13
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: QTcF (msec)
Arm/Group | BTDS | Placebo
Number analyzed (Participants) | 44 | 44
QTcF (msec)
  QTcF Day 6 | -1.04 (7.32) | -2.33 (8.07)
  QTcF Day 13 | 4.13 (8.30) | -1.88 (7.67)
Statistical Analysis 1: Comparison: BTDS vs Placebo; Day 6 analysis; Test type: Superiority or Other; p = .427, ANCOVA; Mean Difference (Final Values) = 1.29, 90% CI 2-sided [-1.4 to 4.0]
Statistical Analysis 2: Comparison: BTDS vs Placebo; Day 13 analysis; Test type: Superiority or Other; p = .001, ANCOVA; Mean Difference (Final Values) = 6.01, 90% CI 2-sided [3.2 to 8.8]

8. Secondary Outcome: The Average Differences From Baseline Between Moxifloxacin and Placebo by Fridericia's Corrected Interval (QTcF) on Day 6 and Day 13
Description: as for outcome 7
Time Frame: Baseline to Day 6 and Day 13
Population: The full analysis population for ECGs (N = 131) was defined as all subjects who received at least 1 dose of study drug and had at least 1 postdose digital QT/QTc evaluation.
  For the comparison of moxifloxacin to placebo (N = 88), the subjects randomized to BTDS were excluded.
Measure: Least Squares Mean (Standard Deviation); unit: QTcF (msec)
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 44 | 44
QTcF (msec)
  QTcF Day 6 | 4.74 (7.21) | -2.12 (8.07)
  QTcF Day 13 | 2.83 (7.81) | -1.85 (7.67)
Statistical Analysis 1: Comparison: Moxifloxacin vs Placebo; Day 6 analysis; Test type: Superiority or Other; p < .001, ANCOVA; Mean Difference (Final Values) = 6.86, 90% CI 2-sided [4.2 to 9.6]
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo; Day 13 analysis; Test type: Superiority or Other; p = .006, ANCOVA; Mean Difference (Final Values) = 4.68, 90% CI 2-sided [1.9 to 7.4]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) that occurred after the signing of the informed consent up to end of study and 7 days after, discontinuation, or SAEs occurring up to 30 days following the last study visit were followed until the AE resolved or stabilized.
Description: AEs were obtained by spontaneous reports, subject interview, and daily diary.
Arm/Group | BTDS | Placebo | Moxifloxacin
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44 | 1/44
Other Adverse Events (participants affected / at risk) | 43/44 | 31/44 | 12/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTDS (N=44) | Placebo (N=44) | Moxifloxacin (N=44)
Abortion induced NOS (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Systematic and nonsystematic assessment
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BTDS (N=44) | Placebo (N=44) | Moxifloxacin (N=44)
Vision blurred (Eye disorders) | 3 | 0 | 0 — Systematic and nonsystematic assessments.
Abdominal pain NOS (Gastrointestinal disorders) | 2 | 3 | 2 — Systematic and nonsystematic assessments.
Constipation (Gastrointestinal disorders) | 17 | 3 | 0 — Systematic and nonsystematic assessments.
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 0 — Systematic and nonsystematic assessments.
Dyspepsia (Gastrointestinal disorders) | 5 | 0 | 2 — Systematic and nonsystematic assessments.
Flatulence (Gastrointestinal disorders) | 4 | 1 | 0 — Systematic and nonsystematic assessments.
Nausea (Gastrointestinal disorders) | 26 | 4 | 4 — Systematic and nonsystematic assessments.
Vomiting NOS (Gastrointestinal disorders) | 16 | 0 | 2 — Systematic and nonsystematic assessments.
Application site burning (General disorders) | 1 | 4 | 0 — Systematic and nonsystematic assessments.
Application site erythema (General disorders) | 7 | 5 | 0 — Systematic and nonsystematic assessments.
Application site irritation (General disorders) | 0 | 3 | 0 — Systematic and nonsystematic assessments.
Application site pruritus (General disorders) | 10 | 12 | 0 — Systematic and nonsystematic assessments.
Fatigue (General disorders) | 5 | 1 | 0 — Systematic and nonsystematic assessments.
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 — Systematic and nonsystematic assessments.
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0 — Systematic and nonsystematic assessments.
Muscle twitching (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Disturbance in attention (Nervous system disorders) | 4 | 1 | 0
Dizziness (Nervous system disorders) | 15 | 4 | 2
Headache (Nervous system disorders) | 22 | 8 | 2
Paraesthesia (Nervous system disorders) | 4 | 3 | 1
Somnolence (Nervous system disorders) | 6 | 4 | 0
Tremor (Nervous system disorders) | 7 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 4 | 1 | 0
Affect lability (Psychiatric disorders) | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 4 | 1
Urinary retention (Renal and urinary disorders) | 6 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 0
Acne aggravated (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 4 | 1 | 1
Application site paraesthesia (General disorders) | 2 | 1 | 0
Asthenia (General disorders) | 2 | 1 | 1
Rigors (General disorders) | 2 | 0 | 1
Thirst (General disorders) | 1 | 2 | 0
Abrasion NOS (Injury, poisoning and procedural complications) | 2 | 0 | 0
Poisoning NOS (Injury, poisoning and procedural complications) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Appetite decreased NOS (Metabolism and nutrition disorders) | 2 | 2 | 0
Pain in limb (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Bruxism (Psychiatric disorders) | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Sweating increased (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Flushing (Vascular disorders) | 2 | 0 | 1

LIMITATIONS AND CAVEATS:
BUP1011 is a safety study. The comparison of buprenorphine vs placebo on QTc (interval corrected for heart rate) values is the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days